CLINICAL TRIAL: NCT01741974
Title: Double-blinded Placebo-controlled Multicenter Study of Anti-atherosclerotic and Estrogen-like Activity of Karinat in Perimenopausal Women
Brief Title: Study of Anti-atherosclerotic and Estrogen-like Activity of Karinat in Perimenopausal Women
Acronym: PEARS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute for Atherosclerosis Research, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IAR-KT-PERI
Record Dates: First submitted 2012-12-02; First posted 2012-12-05 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-01

CONDITIONS: Menopausal Syndrome; Atherosclerosis
Keywords: perimenopause; phytoestrogen; atherosclerosis; intima-media thickness
MeSH Terms: conditions — Atherosclerosis | interventions — karinat

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Karinat (Active Comparator): Karinat 500 mg tablet by mouth three times a day
  Interventions: Dietary Supplement: Karinat
- Sugar pill (Placebo Comparator): Placebo tablet 500 mg by mouth three times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Karinat
  Arms: Karinat
Drug: Placebo — Sugar pill manufactured to mimic Karinat 500 mg tablet
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to investigate the anti-atherosclerotic and anti-climacteric action of natural drug Karinat based on phytoestrogen-rich botanicals in perimenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Perimenopausal women aged 45 to 60 years with intact womb and ovaries
* The absence of menstruations between 6 to 24 months
* Last menstruation after the age of 40 years
* Follicle-stimulating hormone (FSH) blood level ≥ 35 ng/ml
* Mammography without nodal form of mastopathy or breast cancer signs
* Absence of hypolipidemic therapy or HRT (hormone replacement therapy) during 6 months before the inclusion

Exclusion Criteria:

* Administration of lipid-lowering drugs, and/or HRT, and/or phytoestrogens during 6 month before inclusion
* Personal history or diagnostic of following diseases:

nodal form of mastopathy or breast cancer any cancer except non-melanoma skin cancer stroke or myocardial infarction chronic renal failure II-III chronic hepatic failure II-III liver cirrhosis chronic heart failure IIa-III exacerbation of chronic stomach or duodenal ulcer obesity (BMI >30 kg/m2) alcohol abuse uncontrolled arterial hypertension (systolic blood pressure > 160 mmHg, diastolic blood pressure > 90 mmHg) current cigarette smoking (>10 cigarettes a day) diabetes mellitus deep vein thrombosis or pulmonary embolism

* Individual intolerance of Karinat or major side effects

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 340 (Actual)
Dates: Start 2005-10; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
B-mode ultrasound of carotid arteries | up to 3 years
  Variation of intima-media thickness of common carotid arteries

SECONDARY OUTCOMES:
Measure of serum atherogenicity | up to 3 years
  Change of the ability of serum to induce cholesterol accumulation in cultured cells